CLINICAL TRIAL: NCT06266455
Title: Transforming Health and Resilience Via Individualized Nutrition in Very Preterm Infants for Extrauterine Growth and Development
Brief Title: Individualized Nutrition to Optimize Preterm Infant Growth and Neurodevelopment
Acronym: THRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00000615
Record Dates: First submitted 2023-09-25; First posted 2024-02-20 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Very Preterm Maturity of Infant; Very Low Birth Weight Infant
Keywords: Magnetic Resonance Imaging; Neurodevelopment; Nutrition; Fortification

STUDY DESIGN:
Intervention Model Description: Prospective, randomized-controlled trial comparing the impact of individualized human milk fortification on somatic growth and neurodevelopment in preterm infants randomized to receive one of three nutritional interventions: standardized (control), adjustable, or targeted human milk fortification.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the nutritional interventions, the clinical and research teams will not be blinded to study intervention. The radiologist and research team members performing MRI interpretation, post-acquisition processing, and quantitative analysis will be blinded to study nutritional intervention arm. Similarly, teams performing neurodevelopmental follow-up will also be blinded to study nutritional intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standardized Fortification (Active Comparator): All study participants will undergo feed advancement and fortification with liquid, bovine-based human milk fortifier (HMF) to an assumed human milk content of 24kcal/oz per the Children's National Hospital NICU standardized clinical feeding protocol. The same milk fortification recipes are utilized for mother's own milk (MOM) and donor human milk (DHM). Each infant's growth trajectory is monitored (weight, length, and head circumference) with dietary modifications performed as needed based on growth parameters.
  Growth failure is defined as a decline in weight-for-age z-score by greater than 1 standard deviation (>1 SD) beginning 1 week after reaching goal fortified feeds. For infants who demonstrate growth failure, Step 1 will be to add medium chain triglyceride (MCT) oil. If growth remains sub-optimal, Step 2 will be to add liquid protein.
  Interventions: Dietary Supplement: Standardized Fortification
- Adjustable (Experimental): Adjustable fortification will begin 1 week after tolerating goal feeds of standardized fortification. Blood urea nitrogen (BUN) level as a marker of protein metabolism will be measured weekly, and supplementation with liquid protein will be adjusted as necessary to maintain a goal BUN level between 9-14mmol/dL, up to a maximum assumed protein intake of 4.5 g/kg/day. Liquid protein supplementation will be modified as follows:
  * BUN Level <9 mmol/dL: Increase by 0.5g/kg/day
  * BUN Level 9-14 mmol/dL: No change
  * BUN Level >14 mmol/dL: Decrease by 0.25g/kg/day
  * BUN Level >20 mmol/dL: Hold for 1 week and re-assess
  Growth failure is defined as a decline in weight-for-age z-score by >1 SD beginning 1 week after achieving BUN within goal range from adjustable fortification. For infants who demonstrate growth failure, MCT oil will be added and increased weekly as needed.
  Interventions: Dietary Supplement: Standardized Fortification; Dietary Supplement: Adjustable Fortification
- Targeted (Experimental): Targeted fortification will begin 1 week after tolerating goal feeds of standardized fortification. Additional supplementation with liquid protein and/or MCT oil will be provided based on twice weekly milk analysis using a mid-infrared human milk analyzer in order to meet macronutrient (carbohydrate, protein, lipid) and energy intake goals per pediatric nutrition guidelines (protein 4-4.5g/kg/day, fat 6-8g/kg/day, energy 120-130kcal/kg/day).
  Growth failure is defined as a decline in weight-for-age z-score by >1 SD beginning 1 week after receiving macronutrient and energy intake within goal range from targeted fortification. For infants with growth failure, total energy intake will be increased with additional protein and/or MCT oil supplementation. Energy intake may be increased weekly as needed.
  Interventions: Dietary Supplement: Standardized Fortification; Dietary Supplement: Adjustable Fortification

INTERVENTIONS:
Dietary Supplement: Standardized Fortification — Fortification with liquid, bovine-based HMF to assumed human milk content of 24kcal/oz
Dietary Supplement: Adjustable Fortification — Additional liquid protein supplementation to maintain serum BUN levels within goal range (9-14mmol/dL)
  Arms: Adjustable
Dietary Supplement: Adjustable Fortification — Additional liquid protein and/or MCT oil supplementation to maintain protein, fat, and energy intake within goal range based upon mid-infrared human milk analysis
  Arms: Targeted

SUMMARY:
Human milk has several well-established benefits but does not adequately meet the increased nutritional demands of the growing preterm infant, necessitating additional nutrient supplementation in a process known as fortification. In U.S. neonatal intensive care units (NICUs), human milk is primarily supplemented using standardized fortification, in which a multicomponent fortifier is added to human milk to achieve assumed nutrient content based on standard milk reference values. However, this method does not account for the significant variability in human milk composition or in preterm infant metabolism, and up to half of all very premature infants experience poor growth and malnutrition using current nutritional practices. Poor postnatal growth has adverse implications for the developing preterm brain and long-term neurodevelopment.

Recent advances allow for individualized methods of human milk fortification, including adjustable and targeted fortification. Adjustable fortification uses laboratory markers of protein metabolism (BUN level) to estimate an infant's protein requirements. In targeted fortification, a milk sample is analyzed to determine its specific macronutrient and energy content, with additional macronutrient supplementation provided as needed to achieve goal values. Emerging data suggest that both methods are safe and effective for improving growth, however information on their comparable efficacy and neurodevelopmental implications are lacking, particularly using advanced quantitative brain MRI (qMRI) techniques.

Through this prospective, randomized-controlled trial, the investigators will compare the impact of individualized human milk fortification on somatic growth and neurodevelopment in preterm infants. Infants will be randomized to receive one of three nutritional interventions: standardized (control group), adjustable, or targeted human milk fortification. Infants will undergo their assigned nutritional intervention until term-equivalent age or discharge home, whichever is achieved first. Brain qMRI will be performed at term-corrected age, and neurodevelopmental follow-up will be performed through 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Birth gestational age (GA) of ≤32 weeks
* Postnatal age ≤4 weeks at time of enrollment
* Maternal plan to provide human milk to infant, and consent to providing donor human milk if insufficient maternal milk supply
* Maternal age > 18 years old

Exclusion Criteria:

* Formula feeding prior to 36 weeks PMA or discharge home (whichever achieved first), either secondary to parental preference or medical necessity
* Dysmorphic features or congenital anomalies suggestive of a genetic syndrome, metabolic disorder, chromosomal abnormality, or congenital infection
* Dysgenetic or major destructive brain lesions detected by head ultrasound before enrollment

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2034-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Weight Gain Velocity | Study enrollment through nutritional intervention endpoint (term-equivalent age (40 weeks PMA [postmenstrual age]) or discharge home, whichever is achieved first)
  Weight gain velocity (grams per kilogram per day)
Length Growth Velocity | Study enrollment through nutritional intervention endpoint (term-equivalent age (40 weeks PMA [postmenstrual age]) or discharge home, whichever is achieved first)
  Length growth velocity (centimeters per week)
Head Circumference Growth Velocity | Study enrollment through nutritional intervention endpoint (term-equivalent age (40 weeks PMA [postmenstrual age]) or discharge home, whichever is achieved first)
  Head circumference growth velocity (centimeters per week)
Total and Regional Brain Volumes | Term-equivalent age (38 to 41 weeks postmenstrual age)
  Total and regional (cortical and deep gray matter, white matter, amygdala-hippocampus, brainstem, cerebellum) brain volumes by MRI
Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) | Term-equivalent age (38 to 41 weeks postmenstrual age)
  Summary scores in 13 different domains (habituation, attention, handling, self-regulation, arousal, excitability, lethargy, hypertonicity, hypotonicity, non-optimal reflex, asymmetric reflex, quality of movement, stress)
Mullen Scales of Early Learning (MSEL) | 18 months corrected age
  Composite score as well as 5 subscores: gross motor, fine motor, visual reception, receptive language, and expressive language (reported as standardized t-scores, higher score indicates a better outcome, mean standardized t-score of 50 with standard deviation of 10)
Mullen Scales of Early Learning (MSEL) | 36 months (3 years) of age
  Composite score as well as 5 subscores: gross motor, fine motor, visual reception, receptive language, and expressive language (reported as standardized t-scores, higher score indicates a better outcome, mean standardized t-score score of 50 with standard deviation of 10)
Wechsler Preschool and Primary Scale of Intelligence (4th edition) (WPPSI-IV) | 60 months (5 years) of age
  Five primary indices: verbal comprehension, visual spatial, working memory, fluid reasoning, and processing speed (higher score indicates better performance, score range 40 to 160)
Differential Abilities Scale (2nd edition)-(DAS-II) | 60 months (5 years) of age
  *For children with significant delays who may be unable to reach basal scores on the WPPSI-IV
  Early years core battery: verbal, nonverbal, and spatial reasoning subtests (higher score indicates better performance, score range 40-170)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No